CLINICAL TRIAL: NCT06695000
Title: A Multi-Site, Randomized, Wait-List Controlled Trial to Assess the Effectiveness and Safety of Digital Cognitive Behavioral Therapy for Insomnia (CBT-I) in Patients with Chronic Insomnia
Brief Title: Digital CBT-I for Chronic Insomnia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: WELT corp (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WCTP-I-C-01
Record Dates: First submitted 2024-11-13; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Insomnia Chronic; Insomnia Disorder
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- digital CBT-I (Experimental)
  Interventions: Device: digital CBT-I
- Waitlist Control (No Intervention)

INTERVENTIONS:
Device: digital CBT-I — The intervention is a digital Cognitive Behavioral Therapy for Insomnia (CBT-I) program, delivered via a mobile application. The program includes structured, self-guided modules focusing on sleep hygiene education, cognitive restructuring, stimulus control, bed time restriction, and relaxation techniques. Each module offers interactive exercises and weekly assignments designed to support behavior change and improve sleep. Participants will receive app-based reminders to encourage regular engagement, with features for tracking progress and adherence throughout the 6 week program.
  Other Names: digital cognitive behavioral therapy for insomnia; SleepQ
  Arms: digital CBT-I

SUMMARY:
This study evaluates the effectiveness and safety of a digital Cognitive Behavioral Therapy program for Insomnia (CBT-I) in individuals with chronic insomnia. Participants will be randomly assigned to either begin digital CBT-I immediately or join a wait-list.

DETAILED DESCRIPTION:
This multi-site, randomized, wait-list controlled trial investigates the effectiveness and safety of a digital Cognitive Behavioral Therapy for Insomnia (CBT-I) program in treating chronic insomnia. Participants will be randomly assigned to start the digital CBT-I immediately or after a wait period. The digital CBT-I program, includes modules on sleep education, cognitive restructuring, stimulus control, sleep restriction, and relaxation techniques. Primary and secondary outcomes will measure insomnia severity, beliefs about sleep, daytime sleepiness, mood, quality of life, productivity, and sleep efficiency. Findings aim to assess the effectiveness of digital CBT-I in improving sleep and daily functioning among chronic insomnia patients in South Korea.

ELIGIBILITY:
Inclusion Criteria:

* Meets diagnostic criteria for insomnia disorder according to the International Classification of Diseases, 10th Revision (ICD-10), including: F51: Nonorganic sleep disorders; G47: Sleep disorders
* Has experienced insomnia symptoms for 3 months or longer.
* Scores 8 or higher on the Insomnia Severity Index (ISI).
* Oral and written fluency in Korean
* Owns a smartphone and is independently able to use apps on a smartphone.
* Voluntarily agrees to participate in this clinical study and provides signed informed consent.

Exclusion Criteria:

* Currently receiving non-pharmacological treatments for insomnia (e.g., CBT-I, light therapy, traditional medicine for sleep) within the past 3 months from screening.
* Diagnosed with other sleep disorders aside from insomnia and currently symptomatic, such as:

  * Obstructive sleep apnea (G47.30)
  * Sleep behavior disorders
  * Restless leg syndrome (G28.8)
  * Narcolepsy (G47.4)
* Has an active, ongoing physical illness that impedes daily functioning, such as:

  * Congestive heart failure
  * Chronic obstructive pulmonary disease (COPD)
  * Acute pain
  * Neurological disorders (e.g., cerebrovascular disease)
  * Neurodegenerative disorders (e.g., dementia, multiple sclerosis)
  * Unstable medical conditions or life expectancy of less than 6 months
* Adjustments in schedule or dosage of sleep medications, antidepressants, anticonvulsants, anxiolytics, or antipsychotics within the past 3 months, or use of PRN (as needed) prescribed sleep medications.
* Engaged in shift work.
* Pregnant individuals or those planning to become pregnant during the study period.
* Any condition that the investigator believes would make participation in the study not in the best interest of the participant or would preclude successful completion of study activities

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Insomnia Severity Index (ISI) Score at Post-Intervention | "From baseline (Visit 1) to post-intervention assessment at 6 weeks
  The Insomnia Severity Index (ISI) measures the severity of insomnia symptoms, with scores ranging from 0 to 28. Higher scores indicate more severe insomnia, with 0-7 representing no clinically significant insomnia, 8-14 mild insomnia, 15-21 moderate insomnia, and 22-28 severe insomnia. This outcome measures the change in ISI score from baseline to 6 weeks, comparing changes between the digital CBT-I group and the waitlist control group.

SECONDARY OUTCOMES:
Change from Baseline in Dysfunctional Beliefs and Attitudes about Sleep (DBAS-16) Score at Post-Intervention (6 Weeks) | From baseline to 6 weeks post-intervention
  The DBAS-16 measures maladaptive beliefs about sleep, with scores ranging from 0 to 160. Higher scores indicate more dysfunctional beliefs. This outcome evaluates the change in DBAS-16 score from baseline to 6 weeks, comparing changes between the digital CBT-I group and the waitlist control group.
Change from Baseline in Epworth Sleepiness Scale (ESS) Score at Post-Intervention (6 Weeks) | From baseline to 6 weeks post-intervention
  The ESS measures daytime sleepiness, with scores ranging from 0 to 24. Higher scores indicate greater sleepiness, with scores above 10 suggesting excessive daytime sleepiness. This outcome assesses the change in ESS score from baseline to 6 weeks
Change from Baseline in Patient Health Questionnaire-9 (PHQ-9) Score at Post-Intervention (6 Weeks) | From baseline to 6 weeks post-intervention
  The PHQ-9 measures the severity of depressive symptoms, with scores ranging from 0 to 27. Higher scores indicate more severe depression, with categories of mild, moderate, moderately severe, and severe depression. This outcome evaluates the change in PHQ-9 score from baseline to 6 weeks, comparing changes between the digital CBT-I group and the waitlist control group.
Change from Baseline in Generalized Anxiety Disorder-7 (GAD-7) Score at Post-Intervention (6 Weeks) | From baseline to 6 weeks post-intervention
  The GAD-7 measures the severity of generalized anxiety symptoms, with scores ranging from 0 to 21. Higher scores indicate greater anxiety, with categories of mild, moderate, and severe anxiety. This outcome assesses the change in GAD-7 score from baseline to 6 weeks, comparing changes between the digital CBT-I group and the waitlist control group.
Change from Baseline in Quality of Life (SF-36) Score at Post-Intervention (6 Weeks) | From baseline to 6 weeks post-intervention
  The SF-36 assesses overall quality of life across multiple domains, with higher scores indicating better quality of life. Scores range from 0 to 100 for each subscale. This outcome measures the change in SF-36 score from baseline to 6 weeks, comparing changes between the digital CBT-I group and the waitlist control group.
Change from Baseline in Work Productivity and Activity Impairment Questionnaire (WPAI-SHP) Score at Post-Intervention (6 Weeks) | From baseline to 6 weeks post-intervention
  The WPAI-SHP assesses work productivity and impairment in daily activities, with scores from 0% to 100%, where higher scores indicate greater impairment. This outcome measures the change in WPAI-SHP score from baseline to 6 weeks, comparing changes between the digital CBT-I group and the waitlist control group.
Change from Baseline in Sleep Efficiency at Post-Intervention (6 Weeks) | From baseline to 6 weeks post-intervention
  Sleep Efficiency (SE) measures the percentage of time spent asleep while in bed, calculated as total sleep time divided by time in bed. Higher values indicate improved sleep efficiency. This outcome assesses the change in SE from baseline to 6 weeks.
Change from Baseline in Sleep Onset Latency at Post-Intervention (6 Weeks) | From baseline to 6 weeks post-intervention
  Sleep Onset Latency (SOL) measures the time (in minutes) it takes to transition from wakefulness to sleep. Lower values indicate improved sleep onset. This outcome assesses the change in SOL from baseline to 6 weeks.
Change from Baseline in Wake After Sleep Onset at Post-Intervention (6 Weeks) | From baseline to 6 weeks post-intervention
  Wake After Sleep Onset (WASO) measures the time (in minutes) spent awake after initially falling asleep until final awakening. Lower values indicate improved sleep continuity. This outcome assesses the change in WASO from baseline to 6 weeks.
Change from Baseline in Total Sleep Time at Post-Intervention (6 Weeks) | From baseline to 6 weeks post-intervention
  Total Sleep Time (TST) measures the total duration of sleep (in minutes) during the night. Higher values indicate improved sleep duration. This outcome assesses the change in TST from baseline to 6 weeks.

OTHER OUTCOMES:
System Usability Scale (SUS) Score for Digital CBT-I at Post-Intervention (6 Weeks) | 6 weeks post-intervention
  The SUS assesses usability of the digital CBT-I intervention, with scores ranging from 0 to 100. Higher scores indicate better usability, with scores above 68 considered above average. This outcome evaluates user experience and satisfaction with the digital CBT-I program.

CONTACTS AND LOCATIONS:
Locations (5):
- South Korea (5):
  - Inje University Ilsan Paik Hospital, Goyang-si, Gyeonggi-do
  - Yongin Severance Hospital, Yongin-si, Gyeonggi-do
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul
  - The Catholic University of Korea, Seoul ST. Mary's Hospital, Seoul, Seoul
  - Ewha Womans University Medical Center, Seoul, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moon DU, Kim J, Sun JH, Lee Y. Applying a mobile intervention for chronic insomnia in routine care: Study protocol for a multicenter randomized controlled trial. Internet Interv. 2025 Jun 20;41:100848. doi: 10.1016/j.invent.2025.100848. eCollection 2025 Sep. PMID 40636932